CLINICAL TRIAL: NCT02316795
Title: Evaluation of Fluorescence Imaging in Sentinel Lymph Node Biopsy for Breast Cancer and Melanoma
Brief Title: Fluorescence Imaging in Sentinel Lymph Node Biopsy for Breast Cancer and Melanoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201302102
Record Dates: First submitted 2014-12-04; First posted 2014-12-15 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Cancer of Breast; Cancer of the Breast; Melanoma; Malignant Melanoma
MeSH Terms: conditions — Breast Neoplasms; Melanoma | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SLN biopsy with ICG injection (Experimental): During the SLN biopsy, the patient will undergo injection of ICG around the breast tumor or melanoma per standard techniques. 1.6 mL of 500 micro-molar ICG will be injected periareolarly (for breast cancer) or peri-tumorly (for melanoma). This will be performed after standard of care technetium-colloid injection. Patients will then undergo the standard SLN biopsy procedure.
  After gamma-probe identification of the SLN, the surgeon will put on the goggle system to attempt to identify the SLN using fluorescence guidance. After this is performed, the goggle system will be removed and the SLN biopsy will be completed per standard techniques. Findings with the goggles will be recorded but will not change how the SLN biopsy is performed.
  Interventions: Procedure: Sentinel lymph node biopsy; Device: Goggle-based device with light-emitting diodes (LED); Drug: Indocynanine Green

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy
  Other Names: SLN biopsy
Device: Goggle-based device with light-emitting diodes (LED)
Drug: Indocynanine Green — This is a infrared fluorescence imaging contrast agent
  Other Names: ICG

SUMMARY:
The NIR light source of our device is based on light-emitting diodes (LEDs), which can deliver sufficient light to biological tissues and induce fluorescence emission to meet the needs of the planned clinical studies. It should be noted that the light source is still well under the US FDA recommended limit for NIR exposure and ANSI standard. In addition, the light source is not laser-based, which is significantly safer than other optical imaging systems utilizing laser technologies. The fluorescence signals will be received by the detector portion of our device. Gain-settings could be easily adjusted during operation to optimize the contrast between high fluorescence areas (tumors) and low fluorescence areas (normal tissues). Real-time fluorescence video will be displayed in the goggle eyepiece as well as on a secondary monitor to facilitate viewing by other surgeons in the room.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with clinically node-negative breast cancer or melanoma being staged with SLN biopsy.
* Negative nodal basin clinical exam.
* At least 18 years of age.
* Able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Contraindications for surgery.
* Receiving any investigational agents.
* History of allergic reactions attributed to ICG or other agents used in the study, including known iodide or seafood allergy.
* Presence of uncontrolled intercurrent illness including, but not limited to, ongoing or active infection of the breast and/or axilla, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant.
* Breastfeeding. Patients who are breastfeeding are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ICG dye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ability for the imaging device to identify the sentinel lymph node (SLN) during the SLN biopsy procedure compared to standard of care gamma-probe identification of the SLN | At the time of the biopsy procedure (approximately 1.5 hours)
  After gamma-probe identification of the SLN, the physician will put on the goggle system to attempt to identify the SLN using fluorescence guidance. After this is performed, the goggle system will be removed and the SLN biopsy will be completed per standard techniques. Findings with the goggles will be recorded but will not change how the SLN biopsy is performed. The surgically-removed SLNs will be pathologically examined under standard protocols.
  Identification of the SLN via fluorescence imaging will be compared to identification of the SLN via standard radiocolloid.
  Fluorescence imaging results will be classified in relation to the "true" status based on the standard SLN biopsy. Descriptive statistics will be utilized to describe the feasibility of the imaging modality in identifying the SLN.
  The main data point collected is "Do ICG-identified node (s) have extra-corporeal gamma activity?"

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Fields, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Liu Y, Akers WJ, Bauer AQ, Mondal S, Gullicksrud K, Sudlow GP, Culver JP, Achilefu S. Intraoperative detection of liver tumors aided by a fluorescence goggle system and multimodal imaging. Analyst. 2013 Apr 21;138(8):2254-7. doi: 10.1039/c3an00165b. PMID 23467534
- [Background] Liu Y, Bauer AQ, Akers WJ, Sudlow G, Liang K, Shen D, Berezin MY, Culver JP, Achilefu S. Hands-free, wireless goggles for near-infrared fluorescence and real-time image-guided surgery. Surgery. 2011 May;149(5):689-98. doi: 10.1016/j.surg.2011.02.007. PMID 21496565
- [Background] Liu Y, Njuguna R, Matthews T, Akers WJ, Sudlow GP, Mondal S, Tang R, Gruev V, Achilefu S. Near-infrared fluorescence goggle system with complementary metal-oxide-semiconductor imaging sensor and see-through display. J Biomed Opt. 2013 Oct;18(10):101303. doi: 10.1117/1.JBO.18.10.101303. PMID 23728180
- [Background] Liu Y, Zhao YM, Akers W, Tang ZY, Fan J, Sun HC, Ye QH, Wang L, Achilefu S. First in-human intraoperative imaging of HCC using the fluorescence goggle system and transarterial delivery of near-infrared fluorescent imaging agent: a pilot study. Transl Res. 2013 Nov;162(5):324-331. doi: 10.1016/j.trsl.2013.05.002. Epub 2013 Jun 5. PMID 23747795
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu